CLINICAL TRIAL: NCT00292929
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Single Intravenous Doses of Artesunate Administered to Healthy Subjects
Brief Title: Study of the Safety of Intravenous Artesunate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: WRAIR 1128; USUHS G183RW; HSRRB A-13276
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2007-03

CONDITIONS: Malaria; Malaria, Cerebral
Keywords: artesunate; artemisinin; falciparum
MeSH Terms: conditions — Malaria; Malaria, Cerebral

INTERVENTIONS:
Drug: Intravenous artesunate

SUMMARY:
The purpose of this study is to establish the safety, tolerability and pharmacokinetics of a single dose of the antimalarial drug artesunate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and non-pregnant, non-lactating females
* Have a normal ECG that may include benign PAC's and PVC's, 1st degree AV block, 2nd degree AV block, Wenckebach
* Have a normal blood pressure (BP) and heart rate (HR). These will be measured after resting supine for about 3 minutes. Normal BP is defined as less than 140 mm Hg systolic and less than 90 mm Hg diastolic. Normal baseline HR is 50 to 90 bpm without symptoms.
* Body mass index between 18 and 29 kg/m**2 or, if out of range, not clinically significant (within 15% of their ideal body weight).
* Be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures
* Have a brief physical examination that demonstrates no clinically significant contraindication for participating in the study.
* If female, have a negative serum pregnancy test at screening and urine pregnancy at admission or be postmenopausal, had a hysterectomy, been sterilized, or agrees to practice effective contraception for the duration fo the study and for a period of 12 weeks after stopping study drug.

Exclusion Criteria:

* Have received any investigational drug or vaccine in the period 0 to 16 weeks before entry to the study.
* Have been on a liquid protein diet in the last year
* Have any clinically significant abnormal physical findings at the screening examination
* Have any clinically significant abnormalities in the results of laboratory screening evaluation
* Have used any prescription drugs within 14 days prior to admission or non-prescription drugs (including herbals or dietary supplements) within 7 days prior to admission
* Existence of any surgical or medical condition that, in the judgement of the clinical investigator, might interfere with the distribution, metabolism or excretion of the drug
* Presence of history of drug allergy requiring treatment. Hay fever is allowed unless it is active or has required treatment within the previous 2 months
* Donation or loss of greater than 400 ml of blood in the period 0 to 12 weeks before entry to the study.
* Serious adverse reaction or hypersensitivity to any drug, particularly artemisinins
* CAGE (screening test for alcoholism) positive (2 out of 4 criteria) or has a history of recent alcohol abuse
* Use of illicit drugs
* Family history of sudden cardiac death or prolonged QT syndrome (defined as 500 msec noted in repeat tracings)
* History of seizure, syncope, or trouble with hearing or balance or other neurological disorder
* History of severe psychiatric disorder or hospitalization for severe psychiatric disorder
* Current job or personal habit of reversed sleep-wake cycle
* History of cardiac disease to include cardiomyopathy, valvular disease, arrhythmia, ischemia, or enlarged heart
* Presence of hepatitis B surface antigen (Hbs-Ag), hepatitis C antibody (antiHCV) or HIV type 1 at screening
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Weina, MD, PhD, Study Director — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States